CLINICAL TRIAL: NCT03512366
Title: Comparative Study Between Desarda and Lichtenstein's Technique for Inguinal Hernia Repair Under Local Anaesthesia: A Double Blind Randomised Controlled Trial
Brief Title: Comparison Between Desarda and Lichtenstein's Technique for Inguinal Hernia Repair Under Local Anaesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, Dr. Prakash Kumar Sasmal, ASSOCIATE PROFESSOR, DEPT. OF GENERAL SURGERY, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IECAIIMSBBSRPGThesis/17-18/38
Record Dates: First submitted 2018-03-14; First posted 2018-04-30 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Hernias Inguinal Reducible; Local Anaesthesia
Keywords: inguinal hernia; lichtenstein's technique; desarda's technique; local anaesthesia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Intervention Model Description: DESARDA'S NO MESH REPAIR:
  It will be performed according to the surgical technique described by Dr. Desarda. A strip will be separated from the upper leaf of the external oblique aponeurosis keeping its insertion and continuity with the muscle intact. This strip will be sutured with the inguinal ligament below and the newly formed upper leaf of EOA above behind the spermatic cord to form the new inguinal floor. Continuous non absorbable prolene 2-0 suture will be used to secure the aponeurotic strip to the inguinal ligament inferiorly , and the strip will be secured superiorly to the internal oblique muscle using interrupted absorbable vicryl sutures. This strip will be put under tension by muscular contraction and works as a shield to prevent recurrence as it gives additional strength to the weakened internal oblique and transverses abdominis muscles.
Who Masked: Participant, Investigator
Masking Description: This will be a double blind trial .The patient will not be revealed about the technique being performed. The investigator who will follow up the patients post operatively in the out-patient clinic will also be blinded about the procedure performed on the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Desarsda's technique (Experimental): These patients wil be operated by the Desarda's technique without using any prosthetic mesh. A strip of external oblique aponeurosis will be used to strengthen the defect.
  Both field block and local infiltration with tumescent anaesthesia techniques will be used for anaesthesia
  Intervention:
  A strip will be separated from the upper leaf of the external oblique aponeurosis keeping its insertion and continuity with the muscle intact. This strip will be sutured with the inguinal ligament below and the muscle arch or conjoint tendon above behind the spermatic cord to form the new inguinal floor. Continuous non absorbable prolene 2-0 suture will be used to secure it to the inguinal ligament inferiorly , and will be secured superiorly to the internal oblique muscle using interrupted absorbable vicryl sutures.
  Interventions: Procedure: Desarda's technique
- Lichtenstein's technique (Active Comparator): These patients will be operated using prosthetic mesh described as Lichtenstein's tension free mesh hernioplasty.
  Both field block and local infiltration with tumescent anaesthesia techniques will be used for anaesthesia.
  Intervention :
  A 6 × 11 cm polypropylene mesh will be fashioned to fit the posterior wall of the inguinal canal and sutured to the fibro-periosteum of the pubic bone and continued laterally, suturing the inferior edge of the mesh to the shelving edge of the inguinal ligament to a point 2 cm lateral to the internal ring. Laterally, 2 cm silt will be made through the mesh to accommodate the cord. while the two tails will be sutured to create a new deep ring made of mesh.
  Interventions: Procedure: Lichtenstein's technique

INTERVENTIONS:
Procedure: Desarda's technique — It will be performed by separating a strip from the upper leaf of the external oblique aponeurosis in continuity with the muscle and suturing it with the inguinal ligament below and the newly formed upper leaf of EOA above behind the spermatic cord to form the new inguinal floor. This strip will be put under tension by muscular contraction and works as a shield to prevent recurrence.
  Other Names: Desarda's No mesh repair
  Arms: Desarsda's technique
Procedure: Lichtenstein's technique — A 6 × 11 cm polypropylene mesh will be fashioned to fit the posterior wall of the inguinal canal and sutured to the fibro-periosteum of the pubic bone and continued laterally, suturing the inferior edge of the mesh to the shelving edge of the inguinal ligament to a point 2 cm lateral to the internal ring.
  Other Names: Lichtenstein's tension free mesh hernioplasty
  Arms: Lichtenstein's technique

SUMMARY:
Inguinal hernia repair is done by two methods. The conventional method uses a prosthetic mesh for strengthening the defect but has been associated with complications. Another new method uses a strip of the external oblique aponeurosis to do the same.There is a necessity to conduct studies comparing the two methods of hernia repair under local anaesthesia in terms of feasibility, economic benefits, faster ambulation with less complications. The purpose of the study is to find a method that will lead to faster disposal of patients and early return to activities, thereby reducing the waiting list of patients that compromises their financial and social spheres and overwhelms the welfare system.

DETAILED DESCRIPTION:
Inguinal hernia is one of the most common treatable surgical conditions. The synthetic prostheses most often used in the inguinal area may in some cases create new clinical problems, such as foreign body sensation in the groin, discomfort, and abdominal wall stiffness, surgical site infections, migration of mesh and may affect procreation and sexual function, The cost and availability of mesh prostheses in smaller towns and underdeveloped regions proves to be a major hindrance. The requirement of the hour is to find a technique that is simple, cost effective, easy to perform, does not require extensive dissection or use of a foreign body, and also gives an acceptable recurrence rate without any major intra or post-operative complications and can be performed as a day care procedure to reduce the burden of cases in our community. A possible option for this is the Desarda method, presented in 2001, which uses an undetached strip of aponeurosis of the external oblique muscle instead of a mesh and has shown to have promising results in studies conducted so far. Several retrospective and randomized controlled trials have shown that local anaesthesia provides the best clinical and economic benefits to patients undergoing inguinal hernia repair. As there have been no studies till date comparing the outcomes for patients operated by these methods under local anaesthesia only, hence this study has been planned to assess if Desarda's technique is suitable to be used as a day care procedure with early return to normal activities after surgery, less post operative discomfort and minimum dose of analgesics and acceptable recurrence rates. This will help reduce the burden of the hospitals as these patients can be operated on a day care basis with minimal discomfort.

ELIGIBILITY:
Inclusion Criteria:

* Primary uncomplicated inguinal hernia
* Male patients aged more than 18 years and less than 80 years
* BMI less than 30kg/sq m
* American Society of Anaesthesiologists (ASA) scale less than III

Exclusion Criteria:

* Patients with recurrent, irreducible or strangulated inguinal hernias
* Patients unable to interpret VAS or give consent
* Patients participating in other clinical trials
* Patients with infection in the inguinal region or epididymo-orchitis
* Patients allergic to local anaesthetics

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients are only included in the trial
Enrollment: 55 (Estimated)
Dates: Start 2017-12-09 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
To compare Desarda and Lichtenstien's inguinal hernia repair techniques under local anaesthesia, in terms of time taken to return to normal gait with comfort post surgery. | 7 days
  Time taken to return to normal gait comfortably after the surgery is calculated based on the ability to walk comfortably or move freely after surgery, as measured by ability to bend, squat, kneel ,stoop.

SECONDARY OUTCOMES:
Time required to return to work | 30 days
  time taken to resume work activities
Early recurrence within 6 months | 6 months
  Appearance of bulge on the operated hernia site is treated as recurrence
Post operative pain | 6 month
  it is assessed on day 8 and 30 using a visual analogue scale. A Visual Analogue Scale is a measurement instrument that tries to measure a characteristic that ranges across a continuum of values and cant easily be directly measured. For ex,amount of pain a patient feels ranges from none to extreme amount of pain. VAS is a straight horizontal line of fixed length, 10 cm used here.It is completed by the patients themselves and helps compare the magnitude of pain at different points of time.
  Here we use a scale from 0 to 10. Patient can choose any number between 0 to 10. For the convenience certain numbers are assigned pictorial depiction of pain facies with description; like : 0- no pain;2- mild, annoying pain;4- nagging, uncomfortable, troublesome pain;6- distressing, miserable pain;8- intense, dreadful, horrible pain;10- worst possible, unbearable, excruciating pain
Presence of wound infection | 6 months
  Collection of purulent material at the site of incision, associated with tenderness, erythema and edema at the incision site, can be associated with systemic signs like fever and leukocytosis. It is evaluated by the investigator based on his clinical acumen and objective evidence of fever and leucocytosis
Presence of seroma | 30 days
  Collection of clear serous fluid pocket at the site of incision as a result of tissue dissection , found on aspiration of fluctuant swelling at wound site or expressed after staple removal. It is evaluated by the investigator based on his clinical acumen.
Presence of haematoma | 30 days
  Localised collection of blood due to vascular injury at the surgical site , found on aspiration of swelling at incision site or expressed after removal of staples.
Loss or change in sensation in the operated groin | 30 days
  sensation of touch over the operated groin compared with the opposite groin to look for hyperaesthesia or allodynia
Foreign body sensation | 6 months
  Patient asked if any perception of a foreign body being implanted in the operated groin is present
Abdominal wall stiffness | 6 months
  Patient is asked to comment if any stiffness is felt in the abdominal wall on the operated side during locomotion or performing day to day activities
Testicular edema/atrophy | 6 months
  Ultrasonography of the scrotum is done pre operatively and after 6 months of the surgery to look for any significant change in size of testes and signs of edema or atrophy

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Prakash Ku Sasmal, MBBS,MS,FNB, Principal Investigator — Associate Professor, Dept. of General Surgery
Locations (1):
- All India Institute of Medical Sciences, Bhubaneswar, Odisha, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Szopinski J, Dabrowiecki S, Pierscinski S, Jackowski M, Jaworski M, Szuflet Z. Desarda versus Lichtenstein technique for primary inguinal hernia treatment: 3-year results of a randomized clinical trial. World J Surg. 2012 May;36(5):984-992. doi: 10.1007/s00268-012-1508-1. PMID 22392354
- [Derived] Sasmal PK, Sahoo A, Mishra TS, Das Poddar KK, Ali SM, Singh PK, Kumar P. Feasibility and outcomes of Desarda vs Lichtenstein hernioplasty by local anesthesia for inguinal hernia: a noninferiority randomized clinical trial. Hernia. 2023 Oct;27(5):1155-1163. doi: 10.1007/s10029-023-02837-5. Epub 2023 Jul 15. PMID 37452974